CLINICAL TRIAL: NCT01195415
Title: Cancer Stem Cells and Inhibition of Hedgehog Pathway Signaling in Advanced Pancreas Cancer: A Pilot Study of GDC-0449 in Combination With Gemcitabine
Brief Title: Vismodegib and Gemcitabine Hydrochloride in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03746; NCI-2011-03746 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UMCC 2010-003 (Other: University of Michigan Comprehensive Cancer Center); 8417 (Other: CTEP); P30CA046592 (NIH); NCT01143415 (obsolete NCT alias)
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Results first posted 2015-10-07 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Recurrent Pancreatic Carcinoma; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vismodegib, gemcitabine hydrochloride) (Experimental): Patients receive vismodegib PO QD on days 1-28 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 (beginning in course 2). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Vismodegib

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This pilot clinical trial studies vismodegib and gemcitabine hydrochloride in treating patients with advanced pancreatic cancer. Vismodegib may stop the growth of pancreatic cancer by blocking blow flow to the tumor. Gemcitabine hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vismodegib and gemcitabine hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain tumor biopsies before and after therapy with GDC-0449 (vismodegib) to evaluate the effect of inhibition of hedgehog signaling on pancreatic cancer stem cells by: evaluating the tumor for number and percentage of pancreatic cancer stem cells before and after treatment with GDC-0449.

SECONDARY OBJECTIVES:

I. To assess progression free survival (PFS) at 3 months following treatment with GDC-0449 and gemcitabine (gemcitabine hydrochloride).

II. To assess response rate to treatment and overall survival in patients with advanced pancreas cancer treated with GDC-0449 alone and in combination with gemcitabine.

III. To evaluate the toxicity of GDC-0449 alone and in combination with gemcitabine.

OUTLINE:

Patients receive vismodegib orally (PO) once daily (QD) on days 1-28 and gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15 (beginning in course 2). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed pancreas cancer
* Patients must have metastatic disease or recurrent disease following surgical therapy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients must have disease accessible for core needle biopsy both prior to initiation of therapy and on day 21 (+ or - 1 day) of GDC-0449 treatment
* No previous systemic therapy for metastatic pancreas cancer is permitted; prior neoadjuvant or adjuvant therapy with chemotherapy and/or radiation is allowed provided that the last day of therapy was at least 6 months prior to registration
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal; < 5 x if liver involved in tumor
* Creatinine < 2.0 mg/dl
* The effects of GDC-0449 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because hedgehog (Hh) signal pathway inhibitors as well as gemcitabine are known to be teratogenic, women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; for appropriate methods of contraception considered acceptable; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately;

  * Pregnancy testing: omen of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL beta-human chorionic gonadotropin [bHCG]) within 10-14 days and within 24 hours prior to the first dose of GDC-0449 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of GDC-0449; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of GDC-0449
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450) may be enrolled with caution; GDC-0449 is a substrate of CYP3A4; however, the in vitro metabolic conversion of GDC-0449 is low; effects of cytochrome (CYP) inducers (e.g., carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St. John's wart, and troglitazone) on clinical concentrations of GDC-0449 are unknown; likewise, the effects of strong inhibitors of CYP3A4 (e.g., clarithromycin, erythromycin, itraconazole, ketoconazole, nefazodone, and telithromycin) on GDC-0449 clinical concentrations are unknown, and caution should be exercised when dosing GDC-0449 concurrently with inhibitors of CYP3A4; in addition, GDC-0449 inhibits CYP2C8, CYP2C9, and CYP2C19 drug metabolism enzymes in vitro at concentrations that may be clinically relevant; therefore, caution should be exercised when dosing GDC-0449 concurrently with medications that are substrates of CYP2C8, CYP2C9, and CYP2C19 and have narrow therapeutic windows
* Ability to understand and willingness to provide written informed consent

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 6 months prior to entering the study or those who have not recovered from adverse events due to agents administered more than 6 months earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449 or other agents used in the study
* Patients on anticoagulation with Coumadin are ineligible; however anticoagulation with enoxaparin is acceptable for study entry
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow capsules
* Patients with clinically active liver disease, including active viral or other hepatitis or cirrhosis, are ineligible
* Patients with uncontrolled hypomagnesemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Patients with > grade 1 hyponatremia or hypocalcemia are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because GDC-0449 is a Hh pathway inhibiting agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with GDC-0449, breastfeeding should be discontinued if the mother is treated with GDC-0449; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with GDC-0449; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2014-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Kim EJ, Sahai V, Abel EV, Griffith KA, Greenson JK, Takebe N, Khan GN, Blau JL, Craig R, Balis UG, Zalupski MM, Simeone DM. Pilot clinical trial of hedgehog pathway inhibitor GDC-0449 (vismodegib) in combination with gemcitabine in patients with metastatic pancreatic adenocarcinoma. Clin Cancer Res. 2014 Dec 1;20(23):5937-5945. doi: 10.1158/1078-0432.CCR-14-1269. Epub 2014 Oct 2. PMID 25278454

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Vismodegib, Gemcitabine Hydrochloride)
Started | 25
Completed | 23
Not Completed | 2
Not completed — No repeat biopsy due to progression | 2

BASELINE CHARACTERISTICS:
Population: Patients treated on protocol.
Arm/Group | Treatment (Vismodegib, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 65 [46 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Median Percent at Baseline and 3 Weeks in CD44+/ CD24+/ ESA+ Cells From Needle Biopsy Calculated Using FACS
Description: The median percentage of CD44+CD24+ESA+ cells from needle biopsy were calculated at baseline and at 3 weeks using FACS. The difference between the two time points was calculated.
Time Frame: 3 weeks
Population: Of the 25 patients enrolled, only 22 were evaluable for the primary endpoint.
Measure: Median (Full Range); unit: percentage of CD44+/ CD24+/ ESA+ cells
Arm/Group | Treatment (Vismodegib, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 22
percentage of CD44+/ CD24+/ ESA+ cells
  Baseline Median % of CD44+/CD24+/ESA+ CSCs | 4.79 [0.43 to 37.2]
  3 Weeks Post Tx Median % of CD44+/CD24+/ESA+ CSCs | 3.09 [0.74 to 45.9]

2. Secondary Outcome: The Number of Participants With an Objective Best Response (CR + PR)
Description: The number of participants with either a complete response (CR) or a partial response (PR) will be calculated. A CR is defined as the disappearance of all target lesions. A PR is defined as at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: Up to 4 weeks
Population: All treated patients were evaluable.
Measure: Number; unit: participants
Arm/Group | Treatment (Vismodegib, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 25
participants | 5

3. Secondary Outcome: Median Progression Free Survival
Description: Median progression free survival was calculated for all treated patients. Assessed using the Kaplan-Meier method. The 95% confidence interval for this estimate will be computed using the Greenwood's formula.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vismodegib, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 25
months | 2.8 [1.4 to 4.7]

4. Secondary Outcome: Percentage of Treated Patients Experiencing Grade 3+ Toxicity Per National Cancer Institute Common Toxicity Criteria (CTC) Version 3.0
Time Frame: Up to 4 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Vismodegib, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 25
percentage of patients | 56

ADVERSE EVENTS:
Arm/Group | Treatment (Vismodegib, Gemcitabine Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 16/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vismodegib, Gemcitabine Hydrochloride) (N=25)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Death (General disorders) | 1 (1) — Death due to disease progression
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vismodegib, Gemcitabine Hydrochloride) (N=25)
Anemia (Blood and lymphatic system disorders) | 17 (29)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Photophobia (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 13 (19)
Ascites (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastroparesis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 14 (16)
Vomiting (Gastrointestinal disorders) | 13 (15)
Chills (General disorders) | 3 (3)
Edema limbs (General disorders) | 7 (8)
Fatigue (General disorders) | 18 (28)
Fever (General disorders) | 10 (14)
General disorders and administration site conditions - Other (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 2 (2)
Papulopustular rash (Infections and infestations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 17 (22)
Aspartate aminotransferase increased (Investigations) | 18 (24)
Blood bilirubin increased (Investigations) | 8 (11)
CD4 lymphocytes decreased (Investigations) | 3 (6)
Creatinine increased (Investigations) | 3 (3)
Lipase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 11 (12)
Neutrophil count decreased (Investigations) | 8 (9)
Platelet count decreased (Investigations) | 13 (18)
Weight gain (Investigations) | 6 (6)
Weight loss (Investigations) | 10 (12)
White blood cell decreased (Investigations) | 10 (13)
Anorexia (Metabolism and nutrition disorders) | 19 (24)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (22)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 13 (17)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 19 (23)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 14 (16)
Headache (Nervous system disorders) | 6 (6)
Somnolence (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 7 (7)
Confusion (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 3 (3)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less